CLINICAL TRIAL: NCT05469165
Title: Blocking the Effects of Serotonin to Prevent Ischemic Mitral Regurgitation: a Randomized Trial (CYPRO-MR)
Brief Title: Serotonin Receptor Blockers in Ischemic Mitral Regurgitation
Acronym: CYPRO-MR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 22229
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Ischemic Mitral Regurgitation
Keywords: Ischemic mitral regurgitation; Myocardial infarction; Mitral valve; Serotonin; Cyproheptadine
MeSH Terms: conditions — Myocardial Infarction | interventions — Cyproheptadine; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyproheptadine 4 Mg Oral Tablet (Experimental): Participants will receive cyproheptadine 4mg tablet orally three times a day for three months, with a daily increase of 4mg/dose if the previous dose was well tolerated, up to 0.5 mg/kg/day.
  Interventions: Drug: Cyproheptadine 4 Mg Oral Tablet
- Placebo (Placebo Comparator): Participants will receive a matched placebo orally three times a day for 3 months. Daily titration similar to the treatment arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cyproheptadine 4 Mg Oral Tablet — Cyproheptadine treatment for 3 months
  Other Names: Cyproheptadine
  Arms: Cyproheptadine 4 Mg Oral Tablet
Other: Placebo — Placebo administration for 3months
  Arms: Placebo

SUMMARY:
This study is intended to investigate the effect of cyproheptadine (a 5HT2B receptor blocker) on mitral regurgitation severity.

DETAILED DESCRIPTION:
Ischemic mitral regurgitation (MR) is a common and morbid complication of myocardial infarction (MI), doubling heart failure and mortality with currently limited therapies. Its mechanisms have been previously linked to left ventricle (LV) remodeling with secondary deformation of otherwise normal mitral leaflets. Recent studies are introducing new mechanistic elements, allowing possibilities for potential pharmacotherapeutic approaches. Normal mitral leaflets have the capacity to enlarge and adapt to even the largest LV dilatation to prevent MR. However, this compensatory mechanism is insufficient after MI, and the leaflets are abnormally thick with fibrotic changes. Those fibrotic changes could be related to a variation in blood serotonin (5-HT) levels after MI, which has been previously reported. Serotonin is a known cause of valve fibrosis through its 5HT type 2B receptor. In sheep models, the investigators have tested the hypothesis that a 5HT type 2B receptor blocker (cyproheptadine) can prevent adverse remodeling in the valve after MI. Cyproheptadine treatment was associated with increased valve leaflet surface, attenuated leaflet thickening and collagen deposition. Importantly, treated animals had less MR compared to non-treated animals.

Thus the present study is a double-blind randomized trial to assess the effect of cyproheptadine on MR severity, mitral valve surface variation, and left ventricular size following MI. Serial imaging (3D echo and MRI) will assess valve adaptation, LV remodeling and MR.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18-80 years old with a 1st episode of STEMI with documented coronary obstruction.
2. Left ventricle ejection fraction (LVEF)<50% and mitral tenting area ≥ 4 cm2, OR LVEF ≤ 40% and inferior/posterior wall motion anomaly, OR LVEF≤30% and wall motion in any territory.

Exclusion Criteria:

1. Inability to provide informed consent
2. Hemodynamic instability / cardiogenic shock / papillary muscle rupture
3. Prior mitral valve procedure/surgery
4. Permanent atrial fibrillation (limiting imaging and MR quantification)
5. Primary mitral disease (endocarditis, rheumatic, degenerative or congenital)
6. More than mild valvular disease (other than mitral) at baseline
7. Planned cardiac surgery (CABG or valve intervention) within 3 months
8. Contraindications for MRI
9. Ongoing treatment with selective serotonin reuptake inhibitor (SSRI)
10. Chronic use of sedative medication
11. Ongoing or planned pregnancy
12. Chronic renal failure with Estimated Glomerular Filtration Rate (eGFR) < 30 mL/min
13. Neurocognitive disorder
14. Symptom or prior episode of urinary obstruction or glaucoma (relative contraindications for cyproheptadine)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in mitral regurgitation severity | Baseline, 3 months
  Incidence of more than mild MR (MRI regurgitant fraction ≥ 20%) at 3 months (measured by MRI)

SECONDARY OUTCOMES:
Change in mitral leaflet size | Baseline, 3 months
  Mitral leaflet size (3D echo) and its variation vs baseline (measured by echocardiography)
Change in mitral regurgitation grade | Baseline, 3 months
  Mitral regurgitation grade (measured by echocardiography). Mitral regurgitation is graded on a scale of I-IV (grade I (mild MR), grade II (moderate MR), grade III (moderate-to-severe MR) and grade IV (severe MR)). A higher mitral regurgitation grade is generally associated with a worse outcome for the patient.
Change in left ventricle size | Baseline, 3 months
  Left ventricle size (measured by MRI )
Change in left ventricle function | Baseline, 3 months
  Left ventricle function (measured by MRI )
Incidence of other valve regurgitation | 3 months
  Incidence of other valve regurgitation (more than mild) (measured by echocardiography)
Change in mitral valve thickness | Baseline, 3 months
  Mitral valve thickness (measured by echocardiography)
Adverse events | 3 months and 1 year
  Composite of: Mortality, Heart failure requiring hospital admission, Mitral valve intervention (surgical/percutaneous)
Ischemic events | 3 months and 1 year
  stroke and myocardial infarction
Bleeding events | 3 months and 1 year
  Bleeding Academic Research Consortium (BARC) definition
Change in weight of participants | Baseline, 3 months
  Weight gain during therapy (self-assessment by participants)
Change in the patient's perception of their health status | Baseline, 3 months
  Self-administered questionnaire : Kansas City Cardiomyopathy Questionnaire (KCCQ). All score are represented on a 0-to-100-point scale (lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life).
Change in the functional capacity of participants | 3 months, 1 year
  6-minutes walk test
Incidence of sedation | Baseline, 3 months
  Incidence of sedation (reported by participants)
Change in depression score | Baseline, 3 months
  Self-administered questionnaire: Patient Health Questionnaire (PHQ-9). The Patient Health Questionnaire has a scale of 0-27, with higher scores indicating a worse outcome for the patient, with more severe depression symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Canada